CLINICAL TRIAL: NCT05546229
Title: Interstitial Fluid Collection Validation Study
Brief Title: Assessment of Methadone and Buprenorphine in Interstitial Fluid
Status: Completed | Type: Observational
Sponsor: Cari Health Inc. (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1332356; 5R44DA044905-03 (NIH)
Record Dates: First submitted 2022-09-15; First posted 2022-09-19 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Opioid Use Disorder
Keywords: methadone; buprenorphine; interstitial fluid
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Controls: Subjects not taking medications for opioid use disorder
  Interventions: Procedure: Microneedle based interstitial fluid collection
- Methadone: Subjects taking methadone for opioid use disorder
  Interventions: Procedure: Microneedle based interstitial fluid collection
- Buprenorphine: Subjects taking buprenorphine for opioid use disorder
  Interventions: Procedure: Microneedle based interstitial fluid collection

INTERVENTIONS:
Procedure: Microneedle based interstitial fluid collection — Interstitial fluid will be collected from the skin using microneedles and suction.

SUMMARY:
The purpose of this research is to determine if common medications for opioid use disorder (i.e., buprenorphine/naloxone, buprenorphine, methadone) and their metabolites (norbuprenorphine [a metabolite of buprenorphine], buprenorphine-3-glucuronide [B3G; a metabolite in buprenorphine], ethylidene dimethyl diphenyl pyrrolidine [EDDP; a metabolite of methadone]) can be detected in the dermal interstitial fluid (i.e., fluid extracted from the surface of the skin). Additional subjects who are not prescribed or taking any of these medications will be included in this study to act as a comparison group

DETAILED DESCRIPTION:
This pilot study is an exploratory feasibility study that aims to determine if common medications for opioid use disorder (OUD; i.e., buprenorphine, methadone) and their metabolites (i.e., norbuprenorphine [a metabolite of buprenorphine], buprenorphine-3-glucuronide [B3G; a metabolite in buprenorphine], ethylidene dimethyl diphenyl pyrrolidine [EDDP; a metabolite for methadone]), can be detected in dermal interstitial fluid (ISF). Microliter volumes of ISF from the surface of the skin will be collected from patients with a prescription for each these medications (buprenorphine n = 10; methadone n = 10) and controls (n=2) using a microneedle patch or minimally invasive microneedle array that may be used in conjunction with a standard vacuum pump. Levels of these medications and their metabolites will then be detected and quantitated in these samples using standard and well-established instrumental analysis for comparison to blood samples.

Aim 1: Detect and quantitate buprenorphine and norbuprenorphine in ISF collected from the surface of the skin using a minimally invasive microneedle array. ISF collected from the surface of the skin will be tested for buprenorphine (i.e., Suboxone®, Subutex®), norbuprenorphine (a metabolite of buprenorphine), and B3G (a metabolite of buprenorphine) using standard instrumental analysis.

Aim 2: Detect and quantitate methadone in ISF collected from the surface of the skin using a minimally invasive microneedle array. ISF collected from the surface of the skin will be tested for methadone and EDDP using standard instrumental analysis.

Aim 3: Establish correspondence between detected medication levels in ISF and blood. Medication levels for buprenorphine and methadone detected in the ISF will be compared to medication levels measured in blood samples for the purpose of understanding the correlation between the ISF and blood levels.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65.
* A prescription for buprenorphine at dose ≥ 16 mg/4mg, a prescription for buprenorphine/naloxone at dose ≥ 16 mg/4mg, a prescription for methadone at dose ≥ 60mg, or part of the control group.
* Taken buprenorphine, buprenorphine/naloxone, or methadone as prescribed in the last 7 days, or part of the control group

Exclusion Criteria:

* A condition preventing or complicating ISF collection. Conditions may include dermatological (skin) condition, immunodeficiency, recent blood donation, anemia, cancer, congestive heart failure, HIV, Hepatitis C [HCV], or tuberculosis [TB].
* Any active severe depression (e.g., suicidal ideation) or mania symptoms.
* Lactation, pregnancy, or intending to become pregnant during the course of the study.
* Alcohol use in the past 7 days.
* Illicit substance use in past 7 days (e.g., heroin, methamphetamines).
* Under a conservatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients receiving medication assisted treatment for opioid use disorder and control subjects not receiving any treatment for this condition.
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Bari, MD, Principal Investigator — Synergy San Diego
Locations (1):
- Synergy San Diego, Lemon Grove, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Cari Health Inc. — http://www.carihealth.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 15 patients recruited. 4 patients not eligible do to screening results that resulted in exclusion based on documented exclusion criteria. 1 extra control recruited instead of expected 2 due to initial 2 controls both of the same sex and the desire to have at least one female and one male control
Period: Overall Study
Arm/Group | Controls | Methadone | Buprenorphine
Started | 3 | 6 | 2
Completed | 3 | 6 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Controls | Methadone | Buprenorphine | Total
Number analyzed (Participants) | 3 | 6 | 2 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 2 | 10
  >=65 years | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 5
  Male | 2 | 4 | 0 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Methadone Concentration in Plasma and Interstitial Fluid (ISF) Before and After Taking a Dose
Description: ISF collected from the surface of the skin along with blood plasma by venipuncture will be tested for methadone using LC-MS analysis.
Time Frame: 1 day
Population: Patients that met the inclusion and exclusion criteria of the study. Only the methadone taking cohort included in this measure. Data collected prior to daily dose of methadone and 3 Hours after taking daily dose of methadone.
Measure: Number; unit: ng/ml
Groups:
- Plasma Level of Methadone Prior to Daily Dose of Methadone: Plasma level of methadone from patient treated with methadone for opioid use disorder: Plasma is collected by venipuncture prior to subject taking their daily dose of greater than or equal to 60 mg methadone.
- Plasma Level of Methadone 3 Hours After Taking Daily Dose: Measure methadone levels in plasma 3 hours after taking daily dose of 60 mg or more of methadone
- Interstitial Fluid Level of Methadone Pre Dose: Measurement of methadone from microneedle-based collection of interstitial fluid prior to daily dose of methadone.
- Interstitial Fluid Level of Methadone 3 Hours After Daily Methadone Dose: Measurement of interstitial fluid level of methadone 3 hours after taking daily dose
Arm/Group | Plasma Level of Methadone Prior to Daily Dose of Methadone | Plasma Level of Methadone 3 Hours After Taking Daily Dose | Interstitial Fluid Level of Methadone Pre Dose | Interstitial Fluid Level of Methadone 3 Hours After Daily Methadone Dose
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng/ml
  Participant A: number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant A | 565 | 640 | 760 | 2000
  Participant B: number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant B | 240 | 441 | 14319 | 17418
  Participant C: number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant C | 96 | 353 | 990 | 1200
  Participant D: number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant D | 330 | 526 | 1700 | 3300
  Participant E: number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant E | 796 | 831 | 4300 | 5800
  Participant F: number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant F | 207 | 382 | 420 | 1300

2. Primary Outcome: Methadone Metabolite/ 2-ethylidene-1, 5-dimethyl-3, 3-diphenylpyrrolidine ( EDDP ) Concentration in ISF and Plasma Before and After Taking a Dose of Methadone
Description: Plasma and ISF collected from the surface of the skin will be tested for methadone metabolite /eddp using LC-MS analysis. Detection will be performed before and 3 hours after taking prescribed dose of methadone.
Time Frame: 1 day
Population: Patients that met the inclusion and exclusion criteria of the study. Only methadone taking cohort included in this measure, including patient taking gabapentin. Data collected prior to daily dose of Methadone and 3 hours after taking daily dose of methadone.
Measure: Number; unit: ng/ml
Groups:
- Plasma EDDP Level Prior to Taking Daily Dose of Methadone: Analyze EDDP in plasma collected by venipucture prior to daily dose of at least 60 mg of methadone. Analyze samples using LC-MS
- Plasma EDDP Level 3 Hours After Taking Daily Dose of Methadone: Analyze EDDP in plasma collected by venipuncture 3 hours after taking daily dose of at least 60 mg of methadone. Analyze samples using LC-MS.
- ISF Levels Prior to Daily Dose: ISF collected by microneedle method and analyzed for EDDP level prior to methadone daily dose.
- ISF Levels 3 Hours After Daily Methadone Dose: ISF collected by microneedle method and analyzed for EDDP level 3 hours after methadone daily dose.
Arm/Group | Plasma EDDP Level Prior to Taking Daily Dose of Methadone | Plasma EDDP Level 3 Hours After Taking Daily Dose of Methadone | ISF Levels Prior to Daily Dose | ISF Levels 3 Hours After Daily Methadone Dose
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng/ml
  Patient A: number analyzed (Participants) | 1 | 1 | 1 | 1
  Patient A | 135 | 137 | 260 | 400
  Patient B: number analyzed (Participants) | 1 | 1 | 1 | 1
  Patient B | 10 | 38 | 290 | 370
  Patient C: number analyzed (Participants) | 1 | 1 | 1 | 1
  Patient C | 21 | 41 | 14 | 62
  Patient D: number analyzed (Participants) | 1 | 1 | 1 | 1
  Patient D | 45 | 40.5 | 0 | 76
  Patient E: number analyzed (Participants) | 1 | 1 | 1 | 1
  Patient E | 54 | 57 | 0 | 280
  Patient F: number analyzed (Participants) | 1 | 1 | 1 | 1
  Patient F | 46 | 74 | 98 | 120

3. Secondary Outcome: Pearson Correlation for Methadone Levels in ISF and Blood
Description: The Pearson correlation coefficient of blood and ISF methadone levels was calculated using the Least Squared Method from Microsoft Excel software.
Time Frame: 1 day
Population: Patients that met the criteria for inclusion and lacked exclusions as per protocol. We also excluded one patient that was taking 800mg of gabapentin qid due to the known effect of gabapentin on methadone clearance and drug-drug interactions. Only methadone taking cohort included in this measure.
Measure: Number; unit: Pearson Correlation Coefficient
Arm/Group | Methadone
Number analyzed (Participants) | 5
Pearson Correlation Coefficient | .805
Statistical Analysis 1: Comparison: Methadone; patient plasma versus isf value for methadone; Test type: Other; p = .0049, t-test, 2 sided; 8 degrees of freedom

4. Secondary Outcome: Pearson Correlation Coefficient for Methadone Metabolite / EDDP Levels in ISF and Blood
Description: The Pearson correlation coefficient between the ISF and blood levels of EDDP were calculated using the Least Squared Method by Microsoft Excel software.
Time Frame: 1 day
Population: Patients that met the criteria for inclusion and lacked exclusions as per protocol. We also excluded one patient that was taking 800mg of gabapentin qid due to the known effect of gabapentin on methadone clearance and drug-drug interactions. Only methadone taking cohort included in this data.
Measure: Number; unit: Pearson Correlation Coefficient
Arm/Group | Methadone
Number analyzed (Participants) | 5
Pearson Correlation Coefficient | .84
Statistical Analysis 1: Comparison: Methadone; Test type: Other; p = .0025, t-test, 2 sided; 8 degrees of freedom

5. Secondary Outcome: Buprenorphine Concentration in Plasma and ISF Before and After a Dose Taken
Description: Plasma collected by venipuncture and ISF collected from the surface of the skin will be tested for buprenorphine using LC-MS analysis before and after a dose of buprenorphine has been taken
Time Frame: 1 day
Population: Patients on 16mg or more of buprenorphine for Opioid Use Disorder. Only the buprenorphine taking cohort included in this outcome measure.
Measure: Number; unit: ng/ml
Groups:
- Plasma Level of Buprenorphine Prior to Taking Daily Dose of Buprenorphine: Plasma is collected immediately prior to ISF collection and prior to daily dose of buprenorphine. Sample is analyzed for buprenorphine using LC-MS.
- Plasma Level of Buprenorphine 3 Hours After Taking Daily Dose of Buprenorphine: Plasma is collected 3 hours after daily dose of buprenorphine. Sample is analyzed for buprenorphine using LC-MS.
- ISF Level of Buprenorphine Before Daily Dose: ISF collected before daily dose of buprenorphine and buprenorphine level analyzed using LC-MS.
- ISF Level of Buprenorphine 3 Hrs After Daily Dose: ISF collected 3 hours after daily dose of buprenorphine and buprenorphine level analyzed using LC-MS.
Arm/Group | Plasma Level of Buprenorphine Prior to Taking Daily Dose of Buprenorphine | Plasma Level of Buprenorphine 3 Hours After Taking Daily Dose of Buprenorphine | ISF Level of Buprenorphine Before Daily Dose | ISF Level of Buprenorphine 3 Hrs After Daily Dose
Number analyzed (Participants) | 2 | 2 | 2 | 2
ng/ml
  Participant G: number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant G | 2339 | 22459 | 6509 | 0
  Participant H: number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant H | 0 | 15663 | 0 | 0

6. Primary Outcome: Methadone and Its Metabolite/ EDDP Concentrations Using Liquid Chromatography Mass Spectroscopy (LC-MS) in Subjects Not Taking Methadone
Description: Plasma collected from subjects not taking methadone by venipuncture and ISF collected from the surface of the skin. Samples tested for methadone and methadone metabolite /eddp using Liquid Chromatography-Mass Spec (LC-MS) analysis .
Time Frame: 1 day
Population: Patients not taking methadone that met the inclusion and exclusion criteria of the study. Includes only control and buprenorphine (BUP) cohorts.
Measure: Number; unit: ng/ml
Groups:
- Methadone Plasma: Collect plasma from subjects not taking methadone and analyze samples for methadone using LC-MS
- Methadone Interstitial Fluid (ISF): Collect ISF samples from subjects that are not taking methadone. Analyze samples for methadone using LC-MS.
- EDDP Plasma: Collect plasma from subjects that are not taking methadone. Analyze samples for EDDP using LC-MS.
- EDDP ISF: Collect ISF from subjects that are not taking methadone. Analyze samples for EDDP using LC-MS.
Arm/Group | Methadone Plasma | Methadone Interstitial Fluid (ISF) | EDDP Plasma | EDDP ISF
Number analyzed (Participants) | 5 | 5 | 5 | 5
ng/ml
  Patient Control 1: number analyzed (Participants) | 1 | 1 | 1 | 1
  Patient Control 1 | 0 | 0 | 0 | 0
  Patient Control 2: number analyzed (Participants) | 1 | 1 | 1 | 1
  Patient Control 2 | 0 | 0 | 0 | 0
  Patient Control 3: number analyzed (Participants) | 1 | 1 | 1 | 1
  Patient Control 3 | 0 | 0 | 0 | 0
  Patient Bup 1: number analyzed (Participants) | 1 | 1 | 1 | 1
  Patient Bup 1 | 0 | 0 | 0 | 0
  Patient Bup 2: number analyzed (Participants) | 1 | 1 | 1 | 1
  Patient Bup 2 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 days after study blood and isf sample collection.
Arm/Group | Controls | Methadone | Buprenorphine
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/6 | 0/2

LIMITATIONS AND CAVEATS:
Difficulty recruiting subjects taking 16 mg or more of buprenorphine. Buprenorphine study group limited to 2 instead of the goal of 10 subjects. Data on buprenorphine reported as area under the curve and reading less than the level of detection for the assay reported as 0. Subject taking gabapentin 800mg 3 times a day was excluded from analysis of the correlation of blood and isf levels due to known drug-drug interaction with methadone.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-08-03): https://cdn.clinicaltrials.gov/large-docs/29/NCT05546229/Prot_001.pdf
  • Informed Consent Form (2022-08-03): https://cdn.clinicaltrials.gov/large-docs/29/NCT05546229/ICF_000.pdf